CLINICAL TRIAL: NCT01846533
Title: Osteoprosis in Type 2 Diabetic Patients- a Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201212080RINC
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes Mellitus; Osteoporosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — CBC/DC & BCS
Oversight: Data Monitoring Committee: No

SUMMARY:
Some possible humoural and cellular mechanism for diabetes related osteoporosis/fractures were proposed and summarzied as the following, (1)Diabetes mellitus increases osteoclast function but decreases osteoblast function, thereby leading to accelerated bone loss, osteopenia and osteoporosis. (2)DM/hyperglycemia induces production of macrophage colony stimulating factor (MCSF), tumor necrosis factor (TNF)-α and receptor activator of nuclear factor-κB ligand (RANKL), all of which are osteoblast-derived activators of osteoclast proliferation and differentiation. (3) DM/hyperglycemia suppresses osteoblast proliferation and function, in part, by decreasing runtrelated transcription factor (Runx)-2, osteocalcin and osteopontin expressions. (4)Adipogenic differentiation of mesenchymal stem cells is increased as indicated by the overexpression of adipocyte differentiation markers, including peroxisome proliferator-activated receptor (PPAR)-g, adipocyte fatty acid binding protein (aP2), adipsin and resistin. A decrease in neovascularization may further aggravate bone loss. (5)Bone quality is also reduced as a result of advanced glycation end products (AGE) production, which may eventually result in low impact or fragility fractures. DM are associated osteoporosis/fracture. The underlying mechanism, especially of type 2 DM, mandates a DM-osteoporosis cohort to elucidate. In clinical practice, to developed preventive strategies from osteoporotic-fracture is also necessary.

DETAILED DESCRIPTION:
It is becoming apparent that both type 1 and type 2 diabetes mellitus are associated with an increased risk for osteoporosis-associated fractures. A meta-analysis by Vestergaard showed that patients with type 1 DM have decreased bone mineral density and increased fracture risk. This study noted a 6.9 relative risk of hip fracture, when the expected relative risk of fracture was only 1.4 based on the BMD. This finding suggests that the increased fracture risk is not entirely accounted for by the lower BMD. It has been demonstrated that the presence of diabetic microvascular complications, including ophthalmic, nephropathic, and neurological, lead to a higher risk of hip fracture in patients with type 1 DM. Unlike patients with type 1 DM, patients with type 2 DM have an average or higher BMD than age-matched controls. However, several studies have demonstrated that patients with type 2 DM have a higher risk of hip, proximal humerus, and foot fractures. Data from the Women's Health Initiative Observational Study indicate that post-menopausal women with diabetes are at an increased risk of hip, foot, and spine fractures, and fractures overall. For a given BMD, diabetic bone appears to be less strong and therefore more likely to fracture. Insulin-like growth factor (IGF)-1, insulin, bone morphogenetic proteins and osteoprotegerin (OPG), serve as anabolic signals to promote bone formation. Among these anabolic mediators, liver-derived IGF-1 is of particular interest since profound growth retardation, small bone size, low BMD and osteoporosis were reported in IGF-1 and IGF-1 receptor deficiencies. Furthermore, insulin was found to directly induce osteogenic action by increasing cell proliferation, differentiation, alkaline phosphatase activity and expression of type Ⅰcollagen and osteocalcin in human osteoblast-like MG-63 cells. Type 1 DM featuring low circulating insulin and IGF-1 levels usually occurs in young children prior to peak bone mass attainment, whereas type 2 DM is common in adults who have already attained peak bone mass.

ELIGIBILITY:
1. inclusion:40-99 years old with type 2 DM patient
2. exclusion:organization people

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: type 2 diabetic patients
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Osteoprosis in type 2 diabetic patients- a cohort study | three years

CONTACTS AND LOCATIONS:
Overall Officials: Kuo Chin Huang, PhD, Principal Investigator — Department of Family Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan